CLINICAL TRIAL: NCT01670201
Title: A Prospective, Open, Non-controlled Clinical Investigation to Evaluate the Adequacy of a New Donor Site Dressing in Surgical Burn Patients.
Brief Title: An Investigation to Evaluate a New Donor Site Dressing in Surgical Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MxT Ag 01
Record Dates: First submitted 2012-06-12; First posted 2012-08-22 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2013-02

CONDITIONS: Donor Site Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mepilex Transfer Ag (Experimental): Mepilex Transfer Ag is a soft silicone wound contact layer that absorbs and transfers exudate, maintains a moist wound healing environment and has antimicrobial properties.
  Interventions: Device: Mepilex Transfer Ag

INTERVENTIONS:
Device: Mepilex Transfer Ag — Silver dressing

SUMMARY:
The investigator will identify the test donor site and test location will be considered on the upper anterior thighs as being the most suitable if available. Circumferential donors will be considered acceptable as well.

Treatment will be initiated in the operation room following debridement and split thickness grafting of wounds. Donors will be harvested at 0.010 - 0.012 in. thickness. Treatment and dressing of test donor site will include hemostasis post harvesting with epinephrine-soaked lap sponges. Once adequate hemostasis is achieved, a Mepilex Transfer Ag dressing will be applied directly to study site. Secondary dressing will include covering with ace wrap.

Healing should be asses after 10-14 days.

DETAILED DESCRIPTION:
A prospective, open, non-controlled clinical investigation to evaluate the adequacy of donor site healing when using a new donor site dressing, Mepilex Transfer Ag approximately 20 subjects from 2 centres in the US, presenting with the need for surgical intervention and grafting for burn injury will be enrolled. Eligible subjects will have a selected donor site designated as a "study site".

ELIGIBILITY:
Inclusion Criteria:

1. Surgical donor sites for deep partial-thickness or full-thickness burns
2. Burn of thermal origin
3. Both genders with an age ≥ 7 years at enrolment
4. Signed informed consent
5. Subjects who are younger than the legal consenting age must in addition to their own assent form have a signature from a legally authorized representative.

Exclusion Criteria:

1. Any known or suspected systemic infection
2. Any known sensitivity to silver or other components/products used in this study.
3. Any active, uncontrolled, progressive or untreated malignancy. A subject who has had a malignant disease in the past, was treated with the expectation of a cure and is currently disease-free, may be considered for study entry.
4. Use of penicillamine, corticosteroid or immunosuppressive medication within 2 months prior to enrollment, or current use of nonsteroidal anti- inflammatory agents which cannot be discontinued, or who is likely to be prescribed these medications or any other medications known to adversely affect wound healing during study participation.
5. Major uncontrolled systemic disorders such as hepatic, renal, neurologic, or endocrinologic disorders.
6. Requires immersion hydrotherapy at any time during study participation (note, showering hydrotherapy is allowed).
7. Subject unwilling to comply with 28 day follow-up.
8. Participation in another investigational study while participating in this study.
9. Bleeding disorders

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Gibran, MD, Principal Investigator — UW Medicine Regional Burn Center Seattle, WA 98104
Locations (2):
- United States (2):
  - LongIsland Plastic Surgical Group, PC, Garden City, New York
  - Harborview Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mepilex Transfer Ag
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mepilex Transfer Ag
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Secondary Outcome: Pain at Dressing Changes
Description: The Medain and Full Range values are presented for all pain scores collected over multiple dressing changes, per participant, over the course of 28 Days.
  Adult ( 13 years and older) patient informed about his/her pain from No pain (0) to Most intense pain (100) imaginable, by using the Visual Analogue Scale ( VAS),
  Children were using the WONG baker faces, they could chose between, no hurt, hurts Little bit, hurts Little more, hurts even more hurts whole lot hurts worst.
Time Frame: 28 days
Measure: Median (Full Range); unit: units on a scale VAS 0-100
Arm/Group | Mepilex Transfer Ag
Number analyzed (Participants) | 8
units on a scale VAS 0-100 | 6.0 [0 to 44]

2. Primary Outcome: Percentage of Participants Who Had > 95 % Epithelialization at Day 10
Time Frame: 10 days
Measure: Number; unit: percentage of participants
Arm/Group | Mepilex Transfer Ag
Number analyzed (Participants) | 8
percentage of participants | 0

ADVERSE EVENTS:
Arm/Group | Mepilex Transfer Ag
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Transfer Ag (N=8)
Worsening disruption of wound healing (Skin and subcutaneous tissue disorders) | 1 (1) — Worsening disruption of wound healing
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Transfer Ag (N=8)
Infection to donor site (Skin and subcutaneous tissue disorders) | 1 (1) — Infection to donor site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less